CLINICAL TRIAL: NCT06554574
Title: A Sequential, Randomized, Double-Blind, Placebo-Controlled, Phase 1, Single and Multiple Ascending Dose Study of LTG-305 Administered Orally to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics in Healthy Male and Female Participants 18 to 55 Years of Age
Brief Title: A Phase 1 Single and Multiple Ascending Dose Study of LTG-305 Administered Orally in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Latigo Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LTG-305-001
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LTG-305 (Experimental)
  Interventions: Drug: LTG-305
- Placebo (Placebo Comparator)
  Interventions: Drug: LTG-305

INTERVENTIONS:
Drug: LTG-305 — Part A: Single-Ascending dose cohorts; Part B: Multiple-ascending dose cohorts

SUMMARY:
This is a sequential, randomized, double-blind, placebo-controlled Phase 1 single (SAD) and multiple (MAD) ascending dose study to evaluate the safety, tolerability, and pharmacokinetics (PK) and Pharmacodynamics of orally administered LTG-305 in healthy male and female participants. The study will also include a randomized, double-blind, placebo-controlled within-participant crossover evaluation of pain tolerance during a cold pressor test in healthy male participants 18-55 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 18 to 55 years, inclusive, at the time of signing the informed consent for SAD and MAD only. For Cold Pressor male participants 18 to 55 years.
* Overtly healthy with no clinically relevant abnormalities based on the medical history, physical examinations, clinical laboratory evaluations, and 12-lead ECG that, in the opinion of the investigator, would affect participant safety.
* Body mass index (BMI) within the range of 18-32 kg/m2 (inclusive).

Exclusion Criteria:

* Clinically significant cardiovascular, hematological, renal, hepatic, pulmonary, endocrine, gastrointestinal, immunological, dermatological, neurological, or psychiatric disease which could interfere with, or the treatment for which might interfere with, the conduct of the study or which would, in the opinion of the investigator, unacceptably increase the participant's risk by participating in the study
* Past or current history or evidence of alcohol abuse and/or dependence on recreational drug use
* Donation of over 500 mL blood ≤ 3 months prior to start of participation
* Participant is under legal custodianship.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single and multiple ascending oral doses of LTG-305 in healthy participants. | Up to 7 or 10 days of dosing
  Incidence, severity, seriousness, and causality of treatment-emergent adverse events (TEAEs)
To evaluate the pharmacodynamics of LTG-305 in healthy male participants. | 0-24 hrs, 1-12 hours
  Change from baseline at various individual time points and at various intervals for time to reach PDT and time to reach PTT, for each dose of LTG-305 vs. placebo.
  Time to reach PDT and time to reach PTT at various individual time points and at various intervals for each dose of LTG-305 vs. placebo.
  Area above the Curve (AAC) calculated via NPRS scores vs. time, for each dose of LTG-305 vs. placebo Exposure response

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Unit, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No